CLINICAL TRIAL: NCT00175448
Title: A Randomized Controlled Trial of Outpatient Physiotherapy Versus a Self-Administered Home Exercise Program Following Discharge Home From Total Hip Arthroplasty
Brief Title: Comparison of Physiotherapy Versus Home Exercise Following Hip Replacement Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Dr. Nelson Greidanus, University of British Columbia
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C02-0249
Record Dates: First submitted 2005-09-11; First posted 2005-09-15 (Estimated); Last update posted 2008-09-25 (Estimated); Status verified 2005-09

CONDITIONS: Arthritis; Arthroscopic Hip Surgery
MeSH Terms: conditions — Arthritis | interventions — Physical Therapy Modalities

INTERVENTIONS:
Procedure: physiotherapy — See Detailed Description.

SUMMARY:
A Randomized Controlled Trial of Outpatient Physiotherapy versus a Self-Administered Home Exercise Program Following Discharge Home from Total Hip Arthroplasty

ELIGIBILITY:
Inclusion Criteria:

* primary THA (cemented or cementless)
* preoperative diagnosis of osteoarthritis (primary or secondary)
* meets objective discharge-to-home test following hip replacement
* ability to speak English and reply to questionnaires written in English
* ability to provide informed consent
* may include patients presenting for their second primary hip arthroplasty

Discharge to Home Criteria

* independent supine-to-sit transfer
* independent sit-to-stand transfer
* walk with walking aid 30 meters
* ascend and descend 3 stairs
* deemed medically fit and safe for home environment by surgeon/nursing/PT

Exclusion Criteria:

* surgery as part of a workers' compensation claim
* arthroplasty performed for trauma or following open reduction and internal fixation, malignancy or inflammatory arthropathy
* intra-operative complication of fracture or sciatic nerve injury
* procedure requiring complex surgical approach other than posterior or anterolateral (ie trochanteric osteotomy/micro 2 incision approach)
* indications for additional primary or revision arthroplasty within the time frame of the study (24 months) in other hip or knee joints which would adversely affect quality of life and functional scores pertaining to the joint of interest

Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2005-09; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Physical function at 16 weeks post THA in patients who received outpatient physiotherapy following discharge home compared to unsupervised self- directed exercises alone (as measured by the WOMAC). | 16 weeks

SECONDARY OUTCOMES:
Does outpatient physiotherapy result in superior outcomes (final outcome) at 1 and 2 years post THA? | 2 years
Does outpatient physiotherapy, compared to a self-directed exercise program, result in greater improvement in:
generic health-related QOL (SF-36) and (HUI3)
pain and stiffness (WOMAC pain and stiffness)
activities of daily living (FSI)
patient satisfaction (Brigham and Women's patient satisfaction)
objective physical function (TUG, Harris Hip, Gait Lab)
What is the marginal cost effectiveness of outpatient physiotherapy versus self-directed exercises?
How does the recovery over time compare between programs (trajectory of recovery) ?
What is the difference in musculoskeletal adverse event rate (ie dislocation)?

CONTACTS AND LOCATIONS:
Overall Officials: Nelson Greidanus, MD, Principal Investigator — University of British Columbia